CLINICAL TRIAL: NCT05103748
Title: Function Evaluation of Older Patients With Vertigo and Intervention Study of New Rehabilitation Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20212067-F-1
Record Dates: First submitted 2021-07-01; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-06

CONDITIONS: Vertigo
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional vestibular rehabilitation (Active Comparator): The patient shook his head horizontally and looked in the direction of head rotation. Repeated 10 times, and then shook his head with eyes closed and repeated 10 times. The patient holds a small visual target to practice. The small visual target is placed about 30cm in front of the patient. The subject moves his head back and forth while keeping his sight on the target.
  Interventions: Behavioral: Traditional vestibular rehabilitation
- Cognitive and vestibular dual task training (Experimental): The patient shook his head horizontally and looked in the direction of head rotation. Repeated 10 times, and then shook his head with eyes closed and repeated 10 times. The patient holds a small visual target to practice. The small visual target is placed about 30cm in front of the patient. The subject moves his head back and forth while keeping his sight on the target. Besides, patients wear headphones to listen to the numbers at the same time. The numbers contain 1 and 2, and they are played randomly. They shake their heads when they hear 1, and nod when they hear 2. The training takes 30 minutes, once a day in the morning and evening.
  Interventions: Behavioral: Cognitive and vestibular dual task training

INTERVENTIONS:
Behavioral: Traditional vestibular rehabilitation — The patient shook his head horizontally and looked in the direction of head rotation. Repeated 10 times, and then shook his head with eyes closed and repeated 10 times. The patient holds a small visual target to practice. The small visual target is placed about 30cm in front of the patient. The subject moves his head back and forth while keeping his sight on the target.
  Arms: Traditional vestibular rehabilitation
Behavioral: Cognitive and vestibular dual task training — The patient shook his head horizontally and looked in the direction of head rotation. Repeated 10 times, and then shook his head with eyes closed and repeated 10 times. The patient holds a small visual target to practice. The small visual target is placed about 30cm in front of the patient. The subject moves his head back and forth while keeping his sight on the target. Besides, patients wear headphones to listen to the numbers at the same time. The numbers contain 1 and 2, and they are played randomly. They shake their heads when they hear 1, and nod when they hear 2. The training takes 30 minutes, once a day in the morning and evening.
  Arms: Cognitive and vestibular dual task training

SUMMARY:
By evaluating the balance, gait and cognitive functions of the elderly patients with vertigo, the relevant functional disorders of the elderly patients with vertigo were clarified, and the functional disorders of the elderly patients with vertigo were improved through the new rehabilitation intervention.

ELIGIBILITY:
Inclusion Criteria:

Older than 60 years old

It meets the diagnostic criteria of vertigo disease

Agree to participate in the experiment

Exclusion Criteria:

Complete paralysis caused by severe cerebrovascular diseases

Patients with disability and dementia and long-term bedridden

Unwilling to cooperate with the visitors

Patients who did not meet the inclusion criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Short physical performance battery scale | 8 weeks
  Each of the three subtests (balance, walking speed and repeated chair sit-to-stand test) of the short physical performance battery scale was scored from 0 to 4. The minimum test score is 0 point and maximum test score is 12 points. Higher scores indicate better physical performance.
Berg balance scale | 8 weeks
  The berg balance scaleis composed of 14 items that assess an individual's performance on specific functional tasks. Each item is scored from 0 to 4. The minimum test score is 0 point and maximum test score is 56 points. Higher scores indicate better balance performance.
Dynamic Gait Index scale | 8 weeks
  Dynamic Gait Index scale consists of 8 items including normal gait on flat ground, gait with speed changes, gait with horizontal head movements, gait with vertical head movements, gait and pivot turn, gait and step over obstacle, gait around obstacles and steps up and down stairs. The performance on each item is rated on a 4-point scale (3, independent walking; 2, mild impairment; 1, moderate impairment; 0, severe disorder). The minimum test score is 0 point and maximum test score is 24 points. Higher scores indicate better gait performance.
Montreal Cognitive Assessment Scale | 8 weeks
  The Montreal Cognitive Assessment Scale includes eight aspects: visuospatial and executive function, nomenclature, memory, attention, language, abstraction, delayed recall, and orientation for a total of 30 points.The score criteria are as follows: ≥26 is considered as normal cognitive function; < 26 is considered as cognitive dysfunction. If the number of years of education ≤12 years, the score is added 1 point to correct cultural influence. The lower the score, the worse the cognitive function.
Dizziness handicap inventory scale | 8 weeks
  The dizziness handicap inventory consists of 25 items divided into 3 domains believed to encompass the impact of the disease: functional (9 questions), emotional (9 questions), and physical (7 questions). Each item is assigned 0, 2, or 4 points; therefore, the dizziness handicap inventory total scores is between 0 and 100 points. Mild dizziness(dizziness handicap inventory scale score ≤30) and moderate to severe dizziness(dizziness handicap inventory scale score >30).
Visual analogue scale | 8 weeks
  The visual analogue scale for dizziness used a straight line of 10 cm in length. The numbers between 0 and 10 were marked at equal intervals along the line. The participants were asked to report their self-perceived dizziness on a visual analogue scale describing the severity of dizziness in everyday life on a continuum from 0 (none dizziness) to 10 (extremely severe dizziness).
Generalized Anxiexy Disorde-7 scale | 8 weeks
  The presence of perceived anxiety was evaluated with the Generalized Anxiety Disorder 7-item scale. A score of≤9 points indicates no or mild anxiety; >9, moderate to severe anxiety.
Morse Fall scale | 8 weeks
  There are six main variables measured by the Morse Fall scale: (1) history of falling (possible score of 0 or 25); (2) secondary diagnosis (0 or 15); (3) ambulatory aid (0, 15, or 30); (4) IV or IV access (0 or 20); (5) gait (0, 10, 20); and (6) mental status (0 or 15). The total score can range from 0-125. The scale developers recommend a cut-off point of 45; though, calibration of the scores for patient symptoms and healthcare setting is advised. In this study setting, Morse Fall scale scores of 0-24 were classified as no risk, 25-50 as low risk and 51-125 as high risk.
Frail scale | 8 weeks
  Frailty was assessed using the frail scale. There are 5 components: fatigue, resistance, ambulation, illnesses, and loss of weight. The presence of each characteristic was scored with 1 point and the absence of each characteristic was scored with 0 point. The frail score ranges from 0 to 5, where a score of 0 represents robust, 1-2 as pre-frail, and 3-5 as frail.
Mini-mental State Examination | 8 weeks
  Mini-mental State Examination includes five aspects: orientation, memory, attention and calculation, recall and language ability, with a total score of 30.The scoring standard is: 27-30 is normal;< 27 was divided into cognitive impairment;Mild cognitive impairment ≥21 and < 27 points;Moderate cognitive impairment 10-20;Severe cognitive impairment ≤9, the higher the score, the better the cognitive function.

SECONDARY OUTCOMES:
Dataset of functional magnetic resonance imaging on brain | 8 weeks
  Dataset of functional magnetic resonance imaging on brain includes functional images, structural images and diffusion tensor images.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Wang, Study Director — Department of Geriatrics, Xijing Hospital, Air Force Medical University
Locations (1):
- The First Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi, China